CLINICAL TRIAL: NCT05830825
Title: The Tether™ - Vertebral Body Tethering System Post-Market Clinical Follow-Up Study in UK
Brief Title: PMCF (Post-Market Clinical Follow-up) Study on The Tether™ in UK (United Kingdom)
Status: Recruiting | Type: Observational
Sponsor: LDR Médical SAS (Industry)
Responsible Party: Sponsor
Organization: Highridge Medical (Industry)
Other Study IDs: SP-PMCF-EU-202301
Record Dates: First submitted 2023-03-30; First posted 2023-04-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Scoliosis Idiopathic
Keywords: Vertebral Body Tethering; Fusionless Spine Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Vertebral Body Tethering (VBT) — Vertebral Body Tethering surgery with the Tether™ in UK
  Other Names: The Tether™ - VBT System

SUMMARY:
The goal of this observational study is to collect information about The Tether™ device in participants with progressive idiopathic scoliosis, Lenke Type 1 curves. The main purpose is to provide assessment of:

* ongoing safety
* probable benefits Participants who will receive The Tether™ during spine surgery will have to attend follow-up visits which are part of standard-of-care.

DETAILED DESCRIPTION:
This study is designed to be prospective. After the initial visit, followed by the surgery, the participant is expected to take part in the study for a time period of 5 years post-surgery.

Patients will be enrolled during a period of 36 months, and the study will last until complete collection of the 5-year follow-up data. Data will be collected at: first follow-up post discharge, 6, 12, 24, 36, 48 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive idiopathic scoliosis;
* Skeletally immature, based on both Risser (<5) and Sanders (<8) assessments;
* Major Cobb angle ≥30° and ≤65°;
* Osseous structure dimensionally adequate to accommodate screw fixation, as determined by radiographic imaging;
* Failed bracing and/or be intolerant to brace wear;
* Lenke Type 1 curves (i.e., main thoracic);
* Signed Informed Consent Form by legal guardian or by the patient if ≥ 16 years old.
* The decision to treat patients with The Tether™ - VBT System was made by the patient's clinician outside of this research

Exclusion Criteria:

* Presence of any systemic infection, local infection, or skin compromise at the surgical site;
* Prior spinal surgery at the level(s) to be treated;
* Known poor bone quality defined as a T-score -1.5 or less;
* Skeletal maturity;
* Any other medical or surgical condition which would preclude the potential benefit of spinal surgery, such as coagulation disorders, allergies to the implant materials, and patients unwillingness or inability to cooperate with post-operative care instructions;
* Unwillingness, inability, or living situation (e.g., custody arrangements, homelessness, detention) that would preclude ability to return to the study site for follow-up visits as described in protocol and Informed Consent;
* Patients who are pregnant at the time of enrollment.

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Skeletally immature patients that require surgical treatment to obtain and maintain correction of progressive idiopathic scoliosis (Lenke Type 1 curves), with a major Cobb angle of 30 to 65 degrees whose osseous structure is dimensionally adequate to accommodate screw fixation, as determined by radiographic imaging. Patients should have failed bracing and/or be intolerant to brace wear.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2033-01-30 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Rate of serious adverse events, and device- and/or procedure-related adverse events | 5 years
  Serious adverse events, and device- and/or procedure-related adverse events (including intra-operative) will be registered at any post-operative time point
Percentage of patients with maintenance of the major Cobb angle ≤ 40 degrees | 60 months post-surgery
  Major Cobb angle will be measured by x-rays

SECONDARY OUTCOMES:
Rate of overall adverse events, relatedness, severity, time to event | 5 years
  Adverse events (including intra-operative) will be registered at any post-operative time point
Rate and types of reoperations | 5 years
  Reoperations will be registered at any post-operative time point
Progression of secondary curves | Pre-operative, first follow-up, 6, 12, 24, 36, 48 and 60 months post-surgery
  Secondary curves will be assessed by x-rays
Development of new curves | First follow-up, 6, 12, 24, 36, 48 and 60 months post-surgery
  New curves development will be assessed by x-rays at each follow-up visit
Device integrity failures | First follow-up, 6, 12, 24, 36, 48 and 60 months post-surgery
  Device integrity will be assessed by x-rays at each follow-up visit
Maintenance/change in Sagittal alignment, lumbar lordosis | Pre-operative, first follow-up, 6, 12, 24, 36, 48 and 60 months post-surgery
  Sagittal alignment and lumbar lordosis will be assessed by x-rays
Patient Reported Outcome Measures (PROMs): Scoliosis Research Society Health-Related Quality of Life Questionnaire (SRS-22r) and EuroQol 5 Dimensions Young (EQ-5D-Y) | Pre-operative, first follow-up, 6, 12, 24, 36, 48 and 60 months post-surgery
  PROMs will be filled in by the participants at each visit. The SRS-22R measures quality of life in 5 domains: function, pain, self-image, mental health, and satisfaction/dissatisfaction. The minimum score in each domain is 1 and maximum is 5. Each item is scored from 1 (the worst) to 5 (the best). The EQ-5D-Y descriptive system will be used to assess the following five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy. Each dimension has 3 levels: no problems, some problems and a lot of problems. The associated Visual Analog Scale (from 0 - the worst health to 100 - the best health) can be used as a quantitative measure of health outcome that reflects the younger patient's own judgement.
Pulmonary function | Pre-operative, 24 and 60 months post-surgery
  Pulmonary function test, using routine spirometry, will be performed at pre-operative, 24 and 60 months post-operative visits
Trunk shape | Pre-operative, first follow-up, 6, 12, 24, 36, 48 and 60 months post-surgery
  Measurements of trunk shape will be collected at pre-operative and each follow-up visit with a standard scoliometer device
Trunk flexibility | Pre-operative, first follow-up, 6, 12, 24, 36, 48 and 60 months post-surgery
  Trunk flexibility will be collected at pre-operative and each follow up visit. Clinical measurements will be done for both forward and lateral bending using the "fingertip- to- floor" method
Spine mobility | Pre-operative, first follow-up, 6, 12, 24, 36, 48 and 60 months post-surgery
  Range of Motion will be evaluated by x-rays pre-operatively and at each follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bernard, MD, Principal Investigator — Saint George's Hospital, London
Locations (3):
- United Kingdom (3):
  - Saint George's Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - University Southampton Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheung ZB, Selverian S, Cho BH, Ball CJ, Kang-Wook Cho S. Idiopathic Scoliosis in Children and Adolescents: Emerging Techniques in Surgical Treatment. World Neurosurg. 2019 Oct;130:e737-e742. doi: 10.1016/j.wneu.2019.06.207. Epub 2019 Jul 5. PMID 31284059
- [Background] El-Hawary R, Chukwunyerenwa C. Update on evaluation and treatment of scoliosis. Pediatr Clin North Am. 2014 Dec;61(6):1223-41. doi: 10.1016/j.pcl.2014.08.007. Epub 2014 Sep 12. PMID 25439021
- [Background] Kikanloo SR, Tarpada SP, Cho W. Etiology of Adolescent Idiopathic Scoliosis: A Literature Review. Asian Spine J. 2019 Jun;13(3):519-526. doi: 10.31616/asj.2018.0096. Epub 2019 Feb 13. PMID 30744305